CLINICAL TRIAL: NCT02605824
Title: Clinical Trial of NAC in Asthma
Acronym: CONA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was closed after we determined that this albuterol/NAC regimen may be associated with excessive bronchoconstriction.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-17919
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — N-monoacetylcystine; Acetylcysteine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20% n-acetylcystine (NAC) (Experimental): NAC (trade name: Mucomyst) is manufactured by American Regent. The active drug studied here is 20% NAC delivered via nebulizer three times per day for seven days.
  Interventions: Drug: n-acetylcystine
- 0.9% saline (Placebo Comparator): Normal saline will be administered as the placebo agent via a nebulizer three times per day for seven days.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: n-acetylcystine — NAC is a mucolytic drug.
  Other Names: Mucomyst; NAC; acetylcystine
  Arms: 20% n-acetylcystine (NAC)
Drug: 0.9% saline — Normal saline is a placebo agent.
  Other Names: Normal saline
  Arms: 0.9% saline

SUMMARY:
This study evaluates 20% n-acetylcystine (NAC) in the treatment of moderate-to-severe asthma that is complicated by mucus in the airway, as determined by CT imaging. The study is a crossover design, which means that half the study participants will get 20% NAC in the first 7-day treatment period and placebo in the next 7-day treatment period; and the other half will get placebo in the first 7-day treatment period and 20% NAC in the next 7-day treatment period.

DETAILED DESCRIPTION:
n-acetylcystine (NAC) is a mucolytic medication, meaning that it breaks apart mucus. Investigators know that mucus is a factor in severe asthma attacks. However, mucus may be a factor in chronic severe asthma as well. This role has been hard to prove because of difficulty in showing that mucus occludes the lumen in chronic severe disease. Using a novel approach of scoring mucus occlusion, investigators have used CT imaging to uncover that a majority of people with severe asthma have at least one lung segment with a mucus plug and 27% have more than four lung segments with mucus plugs.

Historically, studies of mucolytics, like NAC, have not shown benefit in other obstructive lung diseases, like COPD. However, utilizing CT mucus scores as a biomarker, investigators believe that mucolytic treatment may prove useful for those with significant mucus impaction.

This is a randomized, double-blind, placebo-controlled phase 4 study of 20% NAC in patients with asthma who also have evidence of mucus in their lungs as determined by CT imaging. Investigators hypothesize that by treating asthmatics, chosen based on the presence of mucus in the airways, with a mucolytic like NAC, will result in an improvement of lung function.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform reproducible spirometry according to ATS criteria
* Clinical history consistent with moderate to severe asthma for 1 year or greater.
* Post-bronchodilator FEV1 <90% of predicted
* Prescription and daily use of inhaled corticosteroid (ICS) equivalent to 240mcg of beclomethasone or greater and a second asthma controller therapy.
* CT mucus score >3 (determined during the initial screening process, provided the prior two conditions are met)
* Written informed consent obtained from participant and ability for participant to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* History of intolerance to study medications.
* Current use of carbamazepine
* Angina which includes a treatment plan with PRN nitroglycerin or nitrites
* Smoking of tobacco or other recreational inhalants in last year and/or >10 pack-year smoking history
* Current participation in an investigational drug trial Concurrent Medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

REFERENCES:
- [Background] Hays SR, Fahy JV. The role of mucus in fatal asthma. Am J Med. 2003 Jul;115(1):68-9. doi: 10.1016/s0002-9343(03)00260-2. No abstract available. PMID 12867239
- [Background] DUNNILL MS. The pathology of asthma, with special reference to changes in the bronchial mucosa. J Clin Pathol. 1960 Jan;13(1):27-33. doi: 10.1136/jcp.13.1.27. PMID 13818688
- See also: Study Center Website — http://acrc.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 subjects were consented to the study but only one remained eligible to continue to the treatment period after baseline eligibility testing and the run-in period.
Period: Overall Study
Arm/Group | 20% N-acetylcystine (NAC) | 0.9% Saline
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only one subject was enrolled into the intervention, and after taking the first dose of NAC on the first treatment dat, they experienced excessive bronchospasm thus making them ineligible to continue and complete the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20% N-acetylcystine (NAC) | 0.9% Saline | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-bronchodilator FEV1 (L)
Description: This is a measure of forced expiratory volume measured in one second, following the administration of 4 puffs of albuterol. This outcome will compare the change in post-bronchodilator FEV1 (L) both before and after treatment.
Time Frame: 7 days
Population: Only one subject was enrolled into the intervention, and after taking the first dose of NAC, they experienced excessive bronchospasm thus making them ineligible to continue and complete the study.
Arm/Group | 20% N-acetylcystine (NAC) | 0.9% Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change CT Mucus Score
Description: The CT Mucus Score describes the number of segments of the lungs that are impacted by mucus. This outcome will compare the change in CT mucus score both at baseline and following each treatment period.
Time Frame: 7 days
Population: as for outcome 1
Arm/Group | 20% N-acetylcystine (NAC) | 0.9% Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: Our definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definitions.
Arm/Group | 20% N-acetylcystine (NAC) | 0.9% Saline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT02605824/Prot_SAP_000.pdf